CLINICAL TRIAL: NCT04893655
Title: Effect of Dobutamine on Hepatic Blood Flow During Goal-directed Hemodynamic Therapy
Acronym: DOBU whipple
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BC-08919
Record Dates: First submitted 2021-04-30; First posted 2021-05-19 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: General Anesthesia
Keywords: hepatic blood flow; dobutamine; hepatic vascular pressure
MeSH Terms: interventions — Dobutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dobutamine (Experimental): dobutamine infusion will be started at 2mcg/kg/min after min 10 minutes dobutamine infusion will be raised to 5mcg/kg/min
  Interventions: Drug: Dobutamine Hydrochloride

INTERVENTIONS:
Drug: Dobutamine Hydrochloride — dobutamine infusion will be started at 2mcg/kg/min after min 10 minutes dobutamine infusion will be raised to 5mcg/kg/min

SUMMARY:
Maintaining adequate perfusion pressure and oxygen supply is essential for organ survival. Splanchnic hypoperfusion during the perioperative period in abdominal surgery may result in mucosal ischemia with increased permeability of the gut barrier. Additionally, the liver is also sensitive for hypoxemia and hypoperfusion, especially during liver surgery.

Anesthetics (such as propofol or sevoflurane) have a cardiovascular depressant effect, resulting in a reduction of cardiac output (CO). Dobutamine is used to counteract myocardial depressant effect of anesthetics. Additionally, dobutamine is frequently used during abdominal surgery to maintain splanchnic perfusion.

Dobutamine could increase hepatic blood flow (HBF) indirectly by increasing cardiac output or directly by stimulating adrenergic receptors in the splanchnic circulation. The hepatic circulation has a large number of alpha and beta adrenergic receptors and could be sensitive for adrenergic stimulation such as dobutamine. Hence, dobutamine could have a direct effect on the hepatic vasculature.

The aim of the study is to evaluate the effect of dobutamine on hepatic blood flow during goal directed hemodynamic therapy and to distinguish between potential direct and indirect effects.

DETAILED DESCRIPTION:
All patients receive standardized anesthesia care for pancreaticoduodenectomy according to the existing departmental protocol for these interventions.

All patients receive individualized goal-directed hemodynamic therapy based on the transpulmonary thermodilution technique.

At designated times, hemodynamic variables will be recorded. These include :

* Heart rate (bpm)
* Central venous pressure (mmHg)
* Systolic arterial pressure (mmHg)
* Diastolic arterial pressure (mmHg)
* Mean arterial pressure (mmHg)
* Cardiac index (L/min/m2)
* Pulse pressure variation (PPV)
* Stroke volume variation (SVV)

Measurements of hepatic flow and pressure will be performed by the surgeon :

* Hepatic flow : in the hepatic artery (arterial HBF) and portal vein (portal HBF).
* Pressure measurements : in portal vein (PPorta) and caval vein (PCava)

Measurements will be done :

* without inotropic support
* with infusion of dobutamine 2mcg/kg/min
* with infusion of dobutamine 5mcg/kg/min

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years ≤ 80 years (female or male).
* ASA I - II - III.
* Able to comprehend, sign and date the written informed consent document to participate in the clinical trial.
* Patient is scheduled for pancreaticoduodenectomy (Whipple's procedure).

Exclusion Criteria:

* Allergy to the medication dobutamine.
* Renal insufficiency (SCr > 2 mg/dL).
* Severe heart failure (EF < 25%).
* Hemodynamic unstable patients.
* Atrial fibrillation.
* Sinus tachycardia > 100 bpm on pre-operative electrocardiogram.
* Sepsis.
* BMI > 40.
* Severe coagulopathy (INR > 2).
* Thrombocytopenia (< 80 x 103 /mcL).
* End stage liver disease and/or portal hypertension.
* Pregnancy and breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
change in portal and arterial hepatic blood flow during goal-directed hemodynamic therapy with dobutamine | from start anesthesia until end of anesthesia, up to a maximum of 11 hours
  flow measurements with echo probe
Changes in portal vein and caval vein pressures before and after dobutamine infusion | from start anesthesia until end of anesthesia, up to a maximum of 11 hours
  pressure measurements with 25gauge needle

SECONDARY OUTCOMES:
change in systemic hemodynamic measurements :cardiac index, during goal-directed hemodynamic therapy with dobutamine | from start anesthesia until end of anesthesia, up to a maximum of 11 hours
  change in cardiac index (measurements with PiCCO catheter)
change in systemic vascular resistance (SVR), during goal-directed hemodynamic therapy with dobutamine | from start anesthesia until end of anesthesia, up to a maximum of 11 hours
  change in systemic vascular resistance (SVR)
change in portal venous resistance (PVR), during goal-directed hemodynamic therapy with dobutamine | from start anesthesia until end of anesthesia, up to a maximum of 11 hours
  change in portal venous resistance (PVR)
change in systemic hemodynamic measurements :heart rate, during goal-directed hemodynamic therapy with dobutamine | from start anesthesia until end of anesthesia, up to a maximum of 11 hours
  change in heart rate (measurements with PiCCO catheter)
change in systemic hemodynamic measurements :blood pressure, during goal-directed hemodynamic therapy with dobutamine | from start anesthesia until end of anesthesia, up to a maximum of 11 hours
  change in blood pressure (measurements with PiCCO catheter)
change in systemic hemodynamic measurements :central venous pressure, during goal-directed hemodynamic therapy with dobutamine | from start anesthesia until end of anesthesia, up to a maximum of 11 hours
  change in cardiac index (measurements with central line)
change in systemic hemodynamic measurements :pulse pressure variation, during goal-directed hemodynamic therapy with dobutamine | from start anesthesia until end of anesthesia, up to a maximum of 11 hours
  change in pulse pressure variation (measurements with PiCCO catheter)
change in systemic hemodynamic measurements :stroke volume variation, during goal-directed hemodynamic therapy with dobutamine | from start anesthesia until end of anesthesia, up to a maximum of 11 hours
  change in stroke volume variation (measurements with PiCCO catheter)
change in systemic hemodynamic measurements : Systemic Vascular Resistance Index (SVRI), during goal-directed hemodynamic therapy with dobutamine | from start anesthesia until end of anesthesia, up to a maximum of 11 hours
  change in Systemic Vascular Resistance Index (SVRI) (measurements with PiCCO catheter)
change in systemic hemodynamic measurements : Left Ventricular contractility (dPmx), during goal-directed hemodynamic therapy with dobutamine | from start anesthesia until end of anesthesia, up to a maximum of 11 hours
  change in Left Ventricular contractility (dPmx) (measurements with PiCCO catheter)

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen Van Limmen, MD, Principal Investigator — UZ Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No